CLINICAL TRIAL: NCT02426827
Title: A Safety and Feasibility Study of the Use of Cervical Spinal Cord Stimulation for Treatment of Cerebral Vasospasm in Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Cervical Spinal Cord Stimulation in Cerebral Vasospasm
Acronym: SCSinCV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Scott C. Palmer, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-007493
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCS in CV (Experimental)
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation

SUMMARY:
The study is a non-blinded evaluation of the use of cervical spinal cord stimulation (SCS) for treatment of patients with Hunt and Hess grade 1-2 subarachnoid hemorrhage and evidence of cerebral vasospasm.

DETAILED DESCRIPTION:
The study is a non-blinded evaluation of the use of cervical spinal cord stimulation (SCS) for treatment of patients with Hunt and Hess grade 1-2 subarachnoid hemorrhage and evidence of cerebral vasospasm. Stimulation will be provided with electrodes placed percutaneously in the upper cervical epidural space. The outcome of 5 patients will be studied with focus on possible adverse events related to the intervention. Vasospasm response to treatment will be measured as a secondary outcome. Middle cerebral artery flow velocity will be followed by transcranial Doppler and clinical outcome measured by NIH stroke scale. Flow velocities will be monitored daily by transcranial Doppler and NIH stroke scale performed daily for 7 days, after which spinal cord stimulation will be discontinued and the epidural lead removed.

ELIGIBILITY:
Inclusion Criteria:

* a history of aneurysmal subarachnoid hemorrhage and will have aneurysm secured by clipping or coiling.
* evidence of vasospasm on TCD with MCA mean flow velocity >120 cm/s.
* Patients must be clinically stable to leave the ICU for the study intervention.
* Patients will have Hunt and Hess grade 1-2 non-traumatic subarachnoid hemorrhage.
* Patient should be oriented patients able to provide informed consent.

Exclusion Criteria:

* Patients with non-aneurysmal hemorrhage
* Patient with coagulopathy (PTT>40, or INR > 1.2)
* thrombocytopenia (platelets <100 x 103 per mm2).
* Use of anticoagulation or antiplatelet medication within the known clinical effective period of the particular medication.
* allergy to nimodipine.
* History of cervical or thoracic spine surgery.
* Skin infection at site of catheter placement.
* Sepsis. Pregnancy. Age less than 18 or greater than 80. Active diagnosis of cancer or history of metastatic cancer. Presence of cardiac defibrillator. Inability or unwillingness of patient to give informed consent. Patients found to be clinically neurologically unstable, hemodynamically unstable, or suffering from unstable intracranial pressure at the time of assessment for lead placement will not have the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Looking at number of patients without an adverse effect | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Palmer, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- [Background] Goellner E, Slavin KV. Cervical spinal cord stimulation may prevent cerebral vasospasm by modulating sympathetic activity of the superior cervical ganglion at lower cervical spinal level. Med Hypotheses. 2009 Sep;73(3):410-3. doi: 10.1016/j.mehy.2009.01.055. Epub 2009 May 5. PMID 19409714
- [Background] North R, Shipley J, Prager J, Barolat G, Barulich M, Bedder M, Calodney A, Daniels A, Deer T, DeLeon O, Drees S, Fautdch M, Fehrenbach W, Hernandez J, Kloth D, Krames ES, Lubenow T, North R, Osenbach R, Panchal SJ, Sitzman T, Staats P, Tremmel J, Wetzel T, American Academy of Pain Medicine. Practice parameters for the use of spinal cord stimulation in the treatment of chronic neuropathic pain. Pain Med. 2007 Dec;8 Suppl 4:S200-75. doi: 10.1111/j.1526-4637.2007.00388.x. No abstract available. PMID 17995571
- [Background] Hosobuchi Y. Electrical stimulation of the cervical spinal cord increases cerebral blood flow in humans. Appl Neurophysiol. 1985;48(1-6):372-6. doi: 10.1159/000101161. PMID 3879799
- [Background] Hosobuchi Y. Treatment of cerebral ischemia with electrical stimulation of the cervical spinal cord. Pacing Clin Electrophysiol. 1991 Jan;14(1):122-6. doi: 10.1111/j.1540-8159.1991.tb04056.x. PMID 1705326
- [Background] Takanashi Y, Shinonaga M. Spinal cord stimulation for cerebral vasospasm as prophylaxis. Neurol Med Chir (Tokyo). 2000 Jul;40(7):352-6; discussion 356-7. doi: 10.2176/nmc.40.352. PMID 10927901
- [Background] Visocchi M. Neuromodulation of cerebral blood flow by spinal cord electrical stimulation: the role of the Italian school and state of art. J Neurosurg Sci. 2008 Jun;52(2):41-7. PMID 18500217
- [Background] Smith CC, Lin JL, Shokat M, Dosanjh SS, Casthely D. A report of paraparesis following spinal cord stimulator trial, implantation and revision. Pain Physician. 2010 Jul-Aug;13(4):357-63. PMID 20648204
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Pluijms WA, Slangen R, Joosten EA, Kessels AG, Merkies IS, Schaper NC, Faber CG, van Kleef M. Electrical spinal cord stimulation in painful diabetic polyneuropathy, a systematic review on treatment efficacy and safety. Eur J Pain. 2011 Sep;15(8):783-8. doi: 10.1016/j.ejpain.2011.01.010. Epub 2011 Feb 22. PMID 21345703
- [Background] Lysakowski C, Walder B, Costanza MC, Tramer MR. Transcranial Doppler versus angiography in patients with vasospasm due to a ruptured cerebral aneurysm: A systematic review. Stroke. 2001 Oct;32(10):2292-8. doi: 10.1161/hs1001.097108. PMID 11588316